CLINICAL TRIAL: NCT04363385
Title: Cohort of Patients With Covid19: Constitution of Blood Samples Collections With Clinical Characterization
Brief Title: Collection of Biological Samples With Clinical Characterization of Covid-19 Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No more inclusion
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: COVIGENET
Record Dates: First submitted 2020-04-21; First posted 2020-04-27 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Covid-19
Keywords: Blood samples; ADN; ARN; plasma
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Collection of blood samples in a cohort of Covid-19 patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Collection of blood sample (Other)
  Interventions: Biological: Biological test

INTERVENTIONS:
Biological: Biological test — Blood sample

SUMMARY:
Biological collection (blood sample) associated with clinical data from Covid-19 patients

DETAILED DESCRIPTION:
SARS-Cov2 is an emerging respiratory virus in the coronavirus family, responsible of the pandemic since November 2019. France, which has more than 17,000 deaths from the virus, is one of the main outbreaks. As of 16 April 2020, more than 76,000 individuals in France have been hospitalized, corresponding to 69% of confirmed cases (https://www.santepubliquefrance.fr).

Most affected patients have more or less marked clinical signs associating fever, cough, dyspnea, myalgia, anosmia, ageusia, digestive disorders. In some cases, the progression is worse with lung disease of varying severity. Indications for hospitalization are essentially the severe forms of Covid-19 disease, characterized by hypoxemic lung disease.

Risk factors for developing severe Covid-19 disease have been identified already: age, co-morbidity such as diabetes, obesity-overweight or cardiovascular diseases. It is assumed that other host-related factors, including genetics, may contribute to the existence of this phenotypic heterogeneity. At present, these factors are not known.

The objective of this research is to constitute a DNA collection from patients with Covid-19, in order to be able to search for genetic factors modulating the clinical phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COVID-19 confirmed on RT-PCR test or chest scanner
* Any age
* Membership in the general social security system
* Inform consent signed by the patient or by legal representatives for minors

Exclusion Criteria:

* Refusal of the patient or one of the legal representatives

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2020-05-31 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Phenotype/genotype correlation research modulating the severity of Covid-19 disease | Anytime in the period of 10 years
  Clinical aggravation markers (admission in intensive care)

SECONDARY OUTCOMES:
Phenotype/transcriptomic correlation research modulating the severity of Covid-19 disease | Anytime in the period of 10 years
  Severity at the Covid-19 Lung Scanner
Phenotype/biomarker correlation research modulating the severity of Covid-19 disease | Anytime in the period of 10 years
  Severity at the Covid-19 Lung Scanner
Development of clinical-biological scores in the severity of Covid-19 disease | Anytime in the period of 10 years
  Evolution of scanographic lesions or pulmonary ultrasound
Development of predictive imaging scores in the severity of Covid-19 disease | Anytime in the period of 10 years
  Evolution of scanographic lesions or pulmonary ultrasound
Identification of pathophysiological pathways to susceptibility to Covid-19 disease | Anytime in the period of 10 years
  Duration of oxygen therapy, artificial ventilation
Identification of genetic markers for treatment response | Anytime in the period of 10 years
  Genome sequencing
Identification of transcriptomic markers for treatment response | Anytime in the period of 10 years
  Sequencing transcriptome
Identification of proteomic for treatment response | Anytime in the period of 10 years
  Proteomic sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier intercommunal de Créteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No